CLINICAL TRIAL: NCT03347578
Title: Evaluation of Diaphragmatic Displacement With Echography in Patients Undergoing Thoracic Surgery
Brief Title: Diaphragmatic Echography After Thoracic Surgery
Acronym: OLVDD
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Physician, Università degli Studi di Ferrara
Other Study IDs: OLV DD
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Surgery, Thoracic; Respiratory Diaphragm; Complication, Postoperative
MeSH Terms: conditions — Postoperative Complications | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lung cancer surgery: All patients undergoing thoracic surgery for lung cancer either with thoracoscopy or thoracotomy will receive diaphragmatic Ultrasonography 2 and 24 hours after surgery
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Diaphragmatic ultrasound was performed to investigate diaphragmatic function after thoracic surgery

SUMMARY:
The investigator evaluated diaphragmatic function in patients undergoing thoracic surgery. Diaphragmatic displacement was evaluated before surgery, 2 and 24 hours after surgery. Also, preoperative spirometry and postoperative spirometry were collected (24 hours after surgery).

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery for lung cancer
* Age > 18
* ASA 2-3

Exclusion Criteria:

* BMI > 35
* Contraindications for epidural catheter positioning
* History of neurodegenerative pathology
* Previous thoracic surgery
* Need for mechanical ventilation after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lung resection surgery for cancer
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic dysfunction | 24 hours after surgery
  Diaphragmatic dysfunction is descripted as a diaphragmatic excursione lower than 10 mm

SECONDARY OUTCOMES:
Postoperative pulmonary complications | 7 days after surgery
  Postoperative pulmonary complications include hypoxemia, severe hypoxemia, bronchospasm, suspected pulmonary infection, new pulmonary infiltrates, atelectasis, pleural effusion

IPD SHARING:
Plan to Share IPD: No